CLINICAL TRIAL: NCT05757440
Title: Efficacy of the Application of the Low-viscosity Resin Infiltration on the Change of Color of the Enamel White Spot Lesions
Brief Title: Effect of Low-viscosity Resin Infiltration on Color Change of Enamel White Spot Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre, Egypt (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20157
Record Dates: First submitted 2023-02-14; First posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-02

CONDITIONS: White Spot Lesion of Tooth
Keywords: Low-viscosity resin infiltration; Icon; color change; white spot enamel lesions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Icon resin (Experimental): Low-viscosity Icon resin infiltration
  Interventions: Other: Icon resin application

INTERVENTIONS:
Other: Icon resin application — Application of the low-viscosity resin infiltration (Icon) to the white spot enamel lesions

SUMMARY:
this study aimed to assess the effect of the application of the low-viscosity Icon resin infiltrate on the color change of the diagnosed white spot enamel lesions (WSLs) over 3-, 6-, and 12-m follow-up periods. The ICDAS scoring system was used to visually diagnose WSLs in a total of 96 anterior teeth in 49 participants and the teeth were then were evaluated for their color change using a spectrophotometer. According to the manufacturer directions the Icon kit was applied to the WSLs-diagnosed teeth as follows: the WSLs were treated with 15% hydrofluoric acid (Icon-Etch) was applied to the lesions for 120 seconds then it was rinsed for 30 seconds. Next, the etched WSLs were treated with 99% ethanol (Icon-dry) and for 30 seconds. Then the Icon-Resin was applied and light cured for 40 seconds. The change of color was done after 3-, 6- and 12-month . The mean and standard deviation values were statistically analyzed with the repeated measure ANOVA test and the Paired sample t-test.

DETAILED DESCRIPTION:
The early caries may not be noticeable till it appears as rough enamel surface that might has chalky-white or even dark spots of brown color with no cavities formed. These spots reported were referred to as the white spot enamel lesions, that can be visually diagnosed with the ICDAS scoring method (International Caries Detection and Assessment System) that was proposed for the assessment of caries including early enamel lesions that are not yet cavitated and appear after through dryness of the enamel surface.

Remineralization of the white spots enamel lesion presents the first choice treatment option. Still it has some short-outcomes, such as the staining-ability and unreliable esthetic results. It was reported that the Icon resin infiltration to masking the white spot enamel lesion at the minute of its application without a detectable change of color up to a period of six months. The Icon resin infiltration technique depends on its low-viscosity that enables its penetration into enamel surface through capillary action, occluding the micro porosities created in the enamel as a result of the white enamel lesions development. So that, the progression of the lesion would be stopped.

Therefore, this clinical study was conducted to assess the effectiveness of the application of the Icon resin infiltration on the change of the color change of the white spot enamel lesions at follow-up periods of 3-, 6-, and 12-months.

ELIGIBILITY:
Inclusion Criteria:

* Age range 14-18 years,
* Good general health,
* Permanent dentition,
* Sound anterior teeth,
* Non-cavitated white spot enamel lesions.

Exclusion Criteria:

* Presence of current orthodontic treatments,
* Presence of retained teeth,
* Presence of congenital or developmental anomalies in the permanent dentition,
* Students having systematic conditions,
* Smoking,
* Bad oral hygiene,
* General health problems,
* Missed anterior teeth,
* Carious anterior teeth,
* Intrinsic and extrinsic staining
* Presence of anterior restorations.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 49 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Color change | Immediate after the application of the Icon resin
  Using the intraoral spectrophotometer, which measures the color differences at the specific follow-up periods. The color difference (ΔE) was calculated with the equation: ΔE*Lab= [(ΔL 2) + (Δa 2) + (Δb 2)] ½. Where L* value represents the lightness of an object, The degree of redness and greenness is represented by a* values, while the degree of blue and yellow components of color was determined by b* values. A higher Delta E means more significant color shift.
Color change | At 3 months
  Using the intraoral spectrophotometer, which measures the color differences at the specific follow-up periods. The color difference (ΔE) was calculated with the equation: ΔE*Lab= [(ΔL 2) + (Δa 2) + (Δb 2)] ½. Where L* value represents the lightness of an object, The degree of redness and greenness is represented by a* values, while the degree of blue and yellow components of color was determined by b* values. A higher Delta E means more significant color shift.
Color change | At 6 months
  Using the intraoral spectrophotometer, which measures the color differences at the specific follow-up periods. The color difference (ΔE) was calculated with the equation: ΔE*Lab= [(ΔL 2) + (Δa 2) + (Δb 2)] ½. Where L* value represents the lightness of an object, The degree of redness and greenness is represented by a* values, while the degree of blue and yellow components of color was determined by b* values. A higher Delta E means more significant color shift.
Color change | At 12 months
  Using the intraoral spectrophotometer, which measures the color differences at the specific follow-up periods. The color difference (ΔE) was calculated with the equation: ΔE*Lab= [(ΔL 2) + (Δa 2) + (Δb 2)] ½. Where L* value represents the lightness of an object, The degree of redness and greenness is represented by a* values, while the degree of blue and yellow components of color was determined by b* values. A higher Delta E means more significant color shift.

CONTACTS AND LOCATIONS:
Overall Officials: Lamiaa M Moharam, Assoc Prof., Study Director — National Research Centre, Egypt
Locations (1):
- National Research Centre, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No